CLINICAL TRIAL: NCT00052299
Title: Gemtuzumab Ozogamicin (GO) Combined With Standard Intensive Chemotherapy Versus Standard Intensive Chemotherapy Alone For Induction/Consolidation In Patients 61-75 Years Old With Previously Untreated AML: A Randomized Phase III Trial (AML-17) Of The EORTC-LG and the GIMEMA-ALWP
Brief Title: Chemotherapy With or Without Gemtuzumab Ozogamicin in Treating Older Patients With Acute Myeloid Leukemia
Acronym: AML-17
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-06012; EORTC-06012; AML-17; GIMEMA-AML-17
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia
Keywords: adult acute monocytic leukemia (M5b); adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); untreated adult acute myeloid leukemia; secondary acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities | interventions — Cytarabine; Etoposide; Gemtuzumab; Idarubicin; Mitoxantrone

ARMS (2):
- ARM A (Experimental): GO + MICE for remission induction followed by GO + mini-ICE for consolidation
  Interventions: Drug: cytarabine; Drug: etoposide; Drug: gemtuzumab ozogamicin; Drug: idarubicin; Drug: mitoxantrone hydrochloride
- ARM B (Active Comparator): MICE for remission induction followed by mini-ICE for consolidation
  Interventions: Drug: cytarabine; Drug: etoposide; Drug: idarubicin; Drug: mitoxantrone hydrochloride

INTERVENTIONS:
Drug: cytarabine
Drug: etoposide
Drug: gemtuzumab ozogamicin
  Arms: ARM A
Drug: idarubicin
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known if combining combination chemotherapy with monoclonal antibody therapy will kill more cancer cells.

PURPOSE: Randomized phase III trial to determine the effectiveness of combination chemotherapy with or without gemtuzumab ozogamicin in treating patients who have acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antileukemic activity of standard induction chemotherapy with or without gemtuzumab ozogamicin in elderly patients with previously untreated acute myeloid leukemia.
* Determine the overall survival of patients treated with these regimens.
* Determine the rate of response, disease-free survival, event-free survival, incidence of relapse, and incidence of death of patients treated with these regimens.
* Determine the rate, type, and grade of toxicity of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to age (61-69 vs 70-75), CD33 positivity (less than 5% vs 5-19% vs 20-80% vs more than 80% vs unknown), initial WBC before hydroxyurea administration if needed (less than 30,000/mm^3 vs at least 30,000/mm^3), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I:

  * Induction (phase I): Patients receive gemtuzumab ozogamicin IV over 2 hours on days 1 and 15.
  * Induction (phase II/MICE regimen): Beginning between days 50 and 53, patients receive mitoxantrone IV over 30 minutes on days 1, 3, and 5; etoposide IV over 1 hour on days 1-3; and cytarabine IV continuously on days 1-7. Bone marrow evaluation is performed on day 29. Patients with partial remission (PR) receive a second course of MICE chemotherapy regimen. Patients with complete remission (CR) after 1 or 2 courses of MICE regimen proceed to consolidation therapy. Patients with progressive disease go off therapy.
  * Consolidation: Beginning within 4 weeks of documentation of CR, patients receive gemtuzumab ozogamicin IV over 2 hours on day 0; idarubicin IV on days 1, 3, and 5; etoposide IV over 1 hour on days 1-3; and cytarabine IV continuously on days 1-5. After at least day 30, patients receive a second consolidation course in the absence of disease progression or unacceptable toxicity.
* Arm II:

  * Induction (MICE regimen): Patients receive mitoxantrone, etoposide, and cytarabine as in arm I induction. Bone marrow evaluation is performed on day 29. Patients with PR receive a second course of MICE chemotherapy regimen. Patients with CR after 1 or 2 courses of MICE regimen proceed to consolidation therapy. Patients with progressive disease go off therapy.
  * Consolidation: Patients receive idarubicin, etoposide, and cytarabine as in arm I consolidation.

Patients are followed monthly for 1 year, every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 450 patients (225 per treatment arm) will be accrued for this study within 3.75 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML)

  * Bone marrow blasts at least 20% by bone marrow aspiration or biopsy
  * FAB subtypes M0-M2 and M4-M7

    * No acute promyelocytic leukemia (FAB subtype M3)
* Previously untreated primary or secondary AML, including AML after myelodysplastic syndromes

  * Hydroxyurea and/or corticosteroid therapy for no more than 14 days allowed
* No blast crisis of chronic myelogenous leukemia
* No AML supervening after other myeloproliferative diseases
* No active CNS leukemia

PATIENT CHARACTERISTICS:

Age

* 61 to 75

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC less than 30,000/mm^3 (pretreatment with hydroxyurea for no more than 14 days allowed)

Hepatic

* Bilirubin no greater than 3 times upper limit of normal (ULN)

Renal

* Creatinine no greater than 3 times ULN

Cardiovascular

* No concurrent severe cardiovascular disease
* No arrhythmias requiring chronic treatment
* No congestive heart failure
* No symptomatic ischemic heart disease

Pulmonary

* No severe pulmonary dysfunction (CTC grade 3-4)

Other

* HIV negative
* No other uncontrolled infection
* No other concurrent malignant disease
* No severe concurrent neurological or psychiatric disease
* No prior alcohol abuse
* No psychological, familial, sociological, or geographical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent hematopoietic growth factors (filgrastim [G-CSF] or sargramostim [GM-CSF]) except for life-threatening infection due to neutropenia

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior enrollment in this trial

Ages: 61 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2002-09; Primary Completion 2008-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Response (complete remission [CR] or complete remission with incomplete recovery of platelet count [CRp]) rate after induction
Disease-free survival after CR/CRp
Incidence of relapse after CR/CRp
Incidence of death without relapse after CR/CRp
Event-free survival
Toxicity (highest grade) assessed by International Working Group CTC v2.0

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Amadori, MD, Study Chair — Azienda Ospedallera Universitaria - Policlinico Tor Vergata, Roma
Locations (55):
- Austria (2):
  - A. oe. Krankenhaus der Barmherzigen Schwestern Kinderabteilung, Linz
  - Allgemeines Krankenhaus - Universitatskliniken, Vienna
- Belgium (8):
  - AZ Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Hopital de Jolimont, Haine-Saint-Paul
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- France (3):
  - Hopital Edouard Herriot, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hotel Dieu de Paris, Paris
- Germany (3):
  - Klinikum der Albert - Ludwigs - Universitaet Freiburg, Freiburg im Breisgau
  - Ruprecht - Karls - Universitaet Heidelberg, Heidelberg
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
- Italy (33):
  - Universita Degli Studi di Bari, Bari
  - Azienda Ospedaliera Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Sanitaria di Bolzano, Bolzano
  - Ospedale Binaghi, Cagliari
  - Ospedale Oncologico A. Businco, Cagliari
  - Ospedale Ferrarotto, Catania
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Azienda Istituti Ospitalieri, Cremona
  - Universita di Ferrara, Ferrara
  - Ospedale S. Antonio Abate, Gallarate Varese
  - Ospedale San Martino, Genoa
  - Universita degli Studi di Messina, Messina
  - Azienda Ospedaliera Papardo, Messina
  - Ospedale Civile Umberto I, Mestre
  - Azienda Ospedaliera - Universitaria di Modena, Modena
  - Azienda Ospedaliera "A. Cardarelli", Naples
  - Federico II University Medical School, Naples
  - Azienda Ospedaliera Maggiore Della Carita, Novara
  - Azienda Ospedale S. Luigi at University of Torino, Orbassano
  - Azienda Ospedaliera Policlinico Paolo Giaccone, Palermo
  - Ospedale Cervello, Palermo
  - Ospedale La Maddalena - Palermo, Palermo
  - Perugia Regional Cancer Center, Perugia
  - Azienda Ospedale - d "S. Salvatore", Pesaro
  - Ospedale Civile Pescara, Pescara
  - Ospedale Sant' Eugenio, Rome
  - Libero Istituto Universitario Campus Bio-Medico, Rome
  - Universita Degli Studi "La Sapeinza", Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - H. San Giovanni-Addolorata Hospital, Rome
  - Istituto di Ematologia Universita - University di Sassari, Sassari
  - Policlinico G. B. Rossi - Borgo Roma, Verona
  - Ospedale San Bortolo, Vicenza
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Maxima Medisch Centrum - Veldhoven, Veldhoven
- Hospital Escolar San Joao, Porto, Portugal

REFERENCES:
- [Derived] Amadori S, Suciu S, Stasi R, Salih HR, Selleslag D, Muus P, De Fabritiis P, Venditti A, Ho AD, Lubbert M, Thomas X, Latagliata R, Halkes CJ, Falzetti F, Magro D, Guimaraes JE, Berneman Z, Specchia G, Karrasch M, Fazi P, Vignetti M, Willemze R, de Witte T, Marie JP. Sequential combination of gemtuzumab ozogamicin and standard chemotherapy in older patients with newly diagnosed acute myeloid leukemia: results of a randomized phase III trial by the EORTC and GIMEMA consortium (AML-17). J Clin Oncol. 2013 Dec 10;31(35):4424-30. doi: 10.1200/JCO.2013.49.0771. Epub 2013 Oct 14. PMID 24127442